CLINICAL TRIAL: NCT05787990
Title: Time-in-Range (TIR), a Novel Continuous Glucose Monitoring (CGM) Based Measure, to Improve Risk Stratification of Microvascular Complications in Type 2 Diabetes
Brief Title: Time-In-Range Based Risk Stratification of Type 2 Diabetes Microvascular Complications
Acronym: TRACK2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Singapore Eye Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CNIG20nov-0005
Record Dates: First submitted 2023-02-16; First posted 2023-03-28 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes; Diabetes Related Complications; Diabetes; Retinopathy (Manifestation); Diabetes; Neuropathy, Polyneuropathy (Manifestation); Diabetes; Nephropathy (Manifestation)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications; Diabetes Mellitus; Retinal Diseases; Polyneuropathies; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tear Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diabetes Microvascular Complication Tests — Continuous glucose monitoring using Freestyle Libre Pro, Foot examination with monofilament and neurothesiometer, HbA1c and Urine Microalbumin Creatinine Ratio, Corneal confocal microscopy, Fundal photography, Optical coherence tomography, Optical cohere

SUMMARY:
The goal of this observational study is to learn about the role of Time-in-Range to stratify the risk of micro vascular complications in adults with type 2 diabetes. The main questions it aims to answer are:

1. Is a lower Time-in-Range associated with a higher risk of diabetes microvascular complications, independent of HbA1c?
2. Is Time-in-Range lower among sulfonylurea and premixed insulin therapy users compared to non-sulfonylurea and non-premixed insulin therapy users, respectively.

DETAILED DESCRIPTION:
Methods/Approach

Participants: Investigators aim to recruit a maximum of 500 adults with type 2 diabetes on medical therapy with an HbA1c between 6-12%. Pregnant women, people undergoing active cancer therapies, people taking oral or injectable steroids and those with chronic kidney disease on dialysis will be excluded as the glycemic profile and the pathology in these patients are significantly different from a typical adult with type 2 diabetes. Stratified recruitment will aim to achieve a minimum number in the four major therapy classes to ensure a heterogeneous and representative sample.

1. Oral drugs ± basal insulin not using sulfonylureas (50-200)
2. Oral drugs ± basal insulin using sulfonylureas (50-200)
3. Insulin replacement using premixed insulin therapy (50-200)
4. Insulin replacement using basal-bolus insulin therapy (50-200)

Baseline assessment

At baseline, detailed medical history and anthropometry will be collected from the participants, and participants will have their HbA1c measured, and glycaemia characterized using a blinded CGM. Blood and urine (if required) will be collected for HbA1c and Albumin-creatinine ratio, respectively. HbA1c test results, if available within 6 weeks and Urine Microalbumin-Creatinine Ratio, if available within 6 months from the date of recruitment will be deemed sufficient and no further tests will be done as part of the research. Neuropathy will be assessed by a non-invasive foot exam with a 10g monofilament and neurothesiometer.

Ophthalmological Assessment

Intra-ocular pressure assessment to check for Glaucoma, Administration of Mydriatic eye drop to dilate the eyes, Retinal fundus photograph, In-vivo corneal confocal microscopy, optical coherence tomography and tear sample collection will be performed at Singapore Eye Research Institute (SERI). Optical coherence tomography and in-vivo corneal confocal microscopy are novel non-invasive techniques that can quantify the ocular degenerative changes in people with diabetes. Importantly these techniques are sensitive enough to detect changes in retinal layers and corneal nerve fibre densities even before signs of overt diabetes retinopathy. Diabetic corneal neuropathy has been considered as the surrogate marker for diabetic peripheral neuropathy.

Images generated form the ophthalmological examinations will be analysed using proprietary software and the data used to study the relation between glycaemia and diabetes complications.

For tear sample collection a standardized strip of filter paper will be placed in the lower lateral fornix for 5 mins.

Medical history

Demographics, diabetes related history, current and past medical therapy, past history of microvascular and macrovascular complications, associated metabolic diseases, admissions, and historical HbA1c readings up to 10 years before will be collected. The above data, where required will be retrieved either from the participants or from the electronic medical records of Singapore General Hospital.

Quantifying Time-in-Range (TIR) using Continuous glucose monitoring.

TIR will be measured in the eligible subjects by continuous glucose monitoring method using a blinded continuous glucose sensor. Subjects will be blinded to the glucose readings and will wear the sensor for two weeks, after which data from the sensor will be downloaded for analysis. If the glucose sensor falls off before 7 days or is retrieved with less than 7 full days of data, the participant will wear a second and final continuous glucose monitoring sensor to record glycemic data. Participants will also answer a short survey on their experience of wearing the sensor.

CGM Data: The blinded CGM will generate 1344 glucose readings over two weeks per participant (one reading every 15 minutes). This data will be downloaded and analyzed to calculate various glucose parameters, including percentage Time-in-Range. Time-in-Range is calculated as the percentage of readings within the target range of 3.9-10 mmol/L.

Patient reported outcomes: Data regarding the user experience of the continuous glucose monitoring will be collected using a short survey (included in Data collection form). Other diabetes related patient reported outcomes will be collected from the SGH EMR retrospectively and prospectively to study the impact of glycaemia and diabetes complications on diabetes related patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes,
* Age >= 21 years,
* Ability to provide informed consent,
* HbA1c done within 6 months of recruitment between 6-12%

Exclusion Criteria:

* Undergoing active chemotherapy or immunotherapy for cancer
* Currently taking oral or injectable steroids
* Chronic kidney disease on dialysis
* Women who are pregnant or breastfeeding

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be recruited from people with type 2 diabetes attending Singapore General Hospital outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Presence of Diabetes Retinopathy | 10 years
  Based on Fundal Photography grading
Presence of Diabetes Neuropathy | 10 years
  Based on 10g monofilament foot examination
Presence of Diabetes Nephropathy | 10 years
  Urine microalbumin-creatinine ratio in mg/g

SECONDARY OUTCOMES:
Continuous glucose monitoring derived glycemic variables | 14 days
  Time-in-Range (70-180 mg/dl)
Severity of Retinal degenerative changes | 10 years
  Based on Optical coherence tomography
Severity of corneal neuropathy | 10 years
  Based on confocal corneal microscopy
Severity of diabetes peripheral neuropathy | 10 years
  Vibration threshold on neurothesiometer

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Rama Chandran, MD, MRCP(UK), Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore